CLINICAL TRIAL: NCT04646798
Title: Hemiarthroplasty Or Total Elbow Arthroplasty for Unreconstructible Distal Humerus Fractures in the Elderly (HoT Elbow): a Feasibility Study
Brief Title: Hemiarthroplasty Or Total Elbow Arthroplasty in the Elderly.
Acronym: HOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R&D Study No: 2011059
Record Dates: First submitted 2020-11-17; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Distal Humerus Fracture
MeSH Terms: conditions — Humeral Fractures, Distal | interventions — Hemiarthroplasty; Arthroplasty, Replacement, Elbow

STUDY DESIGN:
Intervention Model Description: To assess the feasibility of undertaking a randomised controlled trial of hemiarthroplasty versus total elbow arthroplasty for patients over the age of 65 who have an unreconstructible distal humeral fracture
Who Masked: Outcomes Assessor
Masking Description: Participant and clinician will not be masked. Data outcomes will be assessed by the research team utilising unique study Identifiers only and group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemi Arthroplasty (HA) of the elbow. (Active Comparator): Hemi Arthroplasty (HA) of the elbow, where the surgeon replaces the bottom of the humerus bone at the elbow.
  Interventions: Other: Hemiarthroplasty
- Total Elbow Arthroplasty (TEA). (Active Comparator): Total Elbow Arthroplasty (TEA), where the surgeon fits a new elbow joint replacing damaged parts of the humerus bone and forearm bone that it joins onto.
  Interventions: Other: Total elbow arthroplasty

INTERVENTIONS:
Other: Hemiarthroplasty — standard surgical approaches to repair of fractured elbows
  Arms: Hemi Arthroplasty (HA) of the elbow.
Other: Total elbow arthroplasty — standard surgical approaches to repair of fractured elbows
  Arms: Total Elbow Arthroplasty (TEA).

SUMMARY:
A feasibility study to assess the practicality, and obtain preliminary data to inform, a definitive Randomise Control Trial (RCT) in patients over the age of 65 diagnosed with un-reconstructible distal humeral fractures, to determine if there are differences in functional outcomes between those undergoing a hemiarthroplasty and a total elbow arthroplasty? Over an 18 month recruitment period the investigators will assess recruitment rates and participants willingness to be randomised to one of two routine clinical treatments. During a 1 year routine clinical follow up period (at 3 time points), routinely collected orthopaedic outcome data will be recorded and differences between groups explored.

DETAILED DESCRIPTION:
Comminuted intra-articular distal humerus fractures (DHF) in the elderly population (over 65 years) have long been a treatment dilemma. Fixation of the fracture often results in development of arthritis and is associated with severe arthrofibrosis (stiffness) and pain. As a consequence, it has become standard practice that elderly patients with these injuries are treated with either elbow hemiarthroplasty (HA) or total elbow arthroplasty (TEA). Both allow immediate mobilisation of the affected arm, with good long term pain and range of motion outcomes reported for both implants in a variety of articles. However each implant has its own advantages and disadvantages.

Elbow HA allows full lifting and loading activities to continue in the operated elbow. However, the concern is that the metal articulation on native cartilage may result in wear and pain associated with this resulting in the need for conversion to a total elbow prosthesis. As this is revision surgery it carries additional risks over first time surgery. Secondly the collateral ligaments have to be reattached and this risks instability following the surgery if this fails.

Patients with TEA are required to avoid lifting and loading activities with the affected arm from the point of surgery and this is ongoing. Such activity can result in failure of the implant with bushing wear, or early progression to aseptic loosening. However, with complete resection of cartilage there is no concern of progressive ulna wear or pain and some literature has suggested a better range of motion due to the semi-constrained nature of the implant meaning condyle retention is not required.

To date no study has directly compared the two arthroplasty options for DHF's in elderly patients. Both implants are currently offered in the Royal Devon and Exeter, National Health Service Foundation Trust (RD&E NHS FT), while other trusts locally are known to offer only one approach. This reflect the uncertainty around which treatment may be better: current provision options are based on the operating surgeon's skills and clinical experience.

To address this state of clinical and personal equipoise will require a large, multi-centred, randomised controlled trial of HA vs TEA, for patients over the age of 65 diagnosed with un-reconstructible DHF's. Before this can be considered the investigators need to assess the feasibility of such a study, and obtain preliminary data to inform its development.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or over at time of surgery
* Scheduled for operative repair by TEA or HA if fracture deemed unfixable.
* Willing and able to provide informed consent
* Willing and able to be randomly allocated to one of two surgical options
* Willing and able to return for local routine clinical follow up

Exclusion Criteria:

* Aged under 65 at time of surgery
* Patients unable to independently consent for inclusion for any reason
* Patients who have had previous elbow joint infections
* Patients who will be unable or unlikely to be able to attend for local routine clinical follow-up (e.g. foreign nationals or holidaymakers who will seek follow-up away from our centre).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 1-18 months
  The number of patients willing to be recruited to the study will be presented as a percentage of the number who were approached, as having met the study inclusion criteria, and invited to join the study.

SECONDARY OUTCOMES:
randomisation/retention rates | 1-30 months
  The number of participants randomised to either of the treatment arms will be presented as a percentage of those recruited (randomisation rate). The number of participants completing all stages of the data collection phases will be presented as a percentage of the number of participants randomised and recruited (retention rate).

OTHER OUTCOMES:
Differences in clinical outcomes between groups as measured by the Oxford Elbow Score (OES) . | 30-36 months
  The OES is a short 12-item Patient Recorded Outcome measure specifically designed to assess outcomes of elbow surgery across 3 unidimensional domains: Elbow function, Pain and Social-psychological.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Smith, MBBCH, Study Director — Royal Devon and Exeter National Health Service Foundation trust
Locations (2):
- United Kingdom (2):
  - NIHR Exeter Clinical Research Facility, Exeter, Devon
  - Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon

IPD SHARING:
Plan to Share IPD: No
feasibility study only

REFERENCES:
- [Background] McKee MD, Veillette CJ, Hall JA, Schemitsch EH, Wild LM, McCormack R, Perey B, Goetz T, Zomar M, Moon K, Mandel S, Petit S, Guy P, Leung I. A multicenter, prospective, randomized, controlled trial of open reduction--internal fixation versus total elbow arthroplasty for displaced intra-articular distal humeral fractures in elderly patients. J Shoulder Elbow Surg. 2009 Jan-Feb;18(1):3-12. doi: 10.1016/j.jse.2008.06.005. Epub 2008 Sep 26. PMID 18823799
- [Background] McKee MD, Wilson TL, Winston L, Schemitsch EH, Richards RR. Functional outcome following surgical treatment of intra-articular distal humeral fractures through a posterior approach. J Bone Joint Surg Am. 2000 Dec;82(12):1701-7. doi: 10.2106/00004623-200012000-00003. PMID 11130643
- [Background] O'Driscoll SW. Optimizing stability in distal humeral fracture fixation. J Shoulder Elbow Surg. 2005 Jan-Feb;14(1 Suppl S):186S-194S. doi: 10.1016/j.jse.2004.09.033. PMID 15726080
- [Background] Huang TL, Chiu FY, Chuang TY, Chen TH. The results of open reduction and internal fixation in elderly patients with severe fractures of the distal humerus: a critical analysis of the results. J Trauma. 2005 Jan;58(1):62-9. doi: 10.1097/01.ta.0000154058.20429.9c. PMID 15674152
- [Background] John H, Rosso R, Neff U, Bodoky A, Regazzoni P, Harder F. [Distal humerus fractures in patients over 75 years of age. Long-term results of osteosynthesis]. Helv Chir Acta. 1993 Sep;60(1-2):219-24. German. PMID 8226060
- [Background] Korner J, Lill H, Muller LP, Hessmann M, Kopf K, Goldhahn J, Gonschorek O, Josten C, Rommens PM. Distal humerus fractures in elderly patients: results after open reduction and internal fixation. Osteoporos Int. 2005 Mar;16 Suppl 2:S73-9. doi: 10.1007/s00198-004-1764-5. Epub 2004 Oct 29. PMID 15517186
- [Background] Pereles TR, Koval KJ, Gallagher M, Rosen H. Open reduction and internal fixation of the distal humerus: functional outcome in the elderly. J Trauma. 1997 Oct;43(4):578-84. doi: 10.1097/00005373-199710000-00003. PMID 9356051
- [Background] Srinivasan K, Agarwal M, Matthews SJ, Giannoudis PV. Fractures of the distal humerus in the elderly: is internal fixation the treatment of choice? Clin Orthop Relat Res. 2005 May;(434):222-30. doi: 10.1097/01.blo.0000154010.43568.5b. PMID 15864057
- [Background] Nestorson J, Ekholm C, Etzner M, Adolfsson L. Hemiarthroplasty for irreparable distal humeral fractures: medium-term follow-up of 42 patients. Bone Joint J. 2015 Oct;97-B(10):1377-84. doi: 10.1302/0301-620X.97B10.35421. PMID 26430013
- [Background] Phadnis J, Watts AC, Bain GI. Elbow hemiarthroplasty for the management of distal humeral fractures: current technique, indications and results. Shoulder Elbow. 2016 Jul;8(3):171-83. doi: 10.1177/1758573216640210. Epub 2016 Apr 21. PMID 27583016
- [Background] Egol K, Koval K, Zuckerman J. Handbook of fractures Fifth Edition. Wolters Kluwer Press
- [Background] McKee MD, Jupiter JB. Fractures of the distal humerus. In: Browner B, Jupiter J, Levine A, Trafton P, editors. Skeletal trauma. 3rd ed. Philadelphia: Lippincott; 2002. p. 765-82
- [Derived] Burden EG, Batten TJ, Thomas W, Evans JP, Smith C. Hemiarthroplasty or total elbow arthroplasty for unreconstructible distal humeral fractures in the elderly (hot elbow): A feasibility study. Shoulder Elbow. 2025 Apr;17(2):200-208. doi: 10.1177/17585732241244722. Epub 2024 Apr 17. PMID 39552682